CLINICAL TRIAL: NCT03626142
Title: Assessing the Effectiveness of Psychiatric Interventions on the Inpatient Unit
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Nolan R, Associate Professor, Psychiatrist, Neurologist, Stanford University
Other Study IDs: 45301
Record Dates: First submitted 2018-07-06; First posted 2018-08-10 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Depressive Symptoms; Suicidal Ideation
MeSH Terms: conditions — Depression; Suicidal Ideation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Left DLPFC aTBS stimulation: Patients who have received accelerated theta burst stimulation delivered to the left dorsolateral prefrontal cortex on the inpatient unit at Stanford
- ACC aTBS stimulation: Patients who have received accelerated theta burst stimulation delivered to the anterior cingulate cortex on the inpatient unit at Stanford
- ECT: Patients who have received ECT on the inpatient unit at Stanford

SUMMARY:
This study will monitor the symptoms of patients who have received an intervention on the psychiatric inpatient unit at Stanford hospital up to 6 months after they have received the intervention. Additionally, the acceptability and feasibility of interventions will be assessed using clinician and patient questionnaires.

DETAILED DESCRIPTION:
Once patients have been discharged from hospital they will be contacted weekly for 4 weeks and then every 2 weeks until 6 months post-intervention in order to monitor their symptoms. Participants will be followed up until the end of the study (6 months after the intervention) or until they no longer meet responder criteria (MADRS score>50% of score before they received the intervention) During the follow-ups for the first 8 weeks, the following assessments will be conducted: Montgomery-Åsberg Depression Rating Scale (MADRS) Scale of suicidal ideation (SSI) Hamilton depression rating scale (HAMD-6) Young Mania Rating Scale (YMRS) Pittsburgh insomnia rating scale (PIRS-20) Quick inventory of depressive symptomatology (QIDS) Immediate Mood Scaler (IMS-12) Beck Depression Inventory (BDI-II) C-SSRS self-report short version

Quality of Life Enjoyment and Satisfaction Questionnaire - Short Form (Q-LES-Q-SF) will be collected at one month post-intervention.

If the participant has a psychiatric diagnosis(/es) other than MDD, questionnaires measuring the symptoms associated with the participant's other psychiatric diagnosis/(es) will also be administered.

Follow-up assessments from 10-24 weeks will include:

MADRS SSI BDI-II C-SSRS self-report short version

If the participant has a psychiatric diagnosis other than MDD, questionnaires measuring the symptoms associated with the participant's other psychiatric diagnosis/(es) will also be administered.

The questionnaires that will be used to assess symptoms associated with primary psychiatric diagnoses are:

* Bipolar disorder: YMRS
* Schizoaffective disorder/ Schizophrenia/Schizophreniform disorder: positive and negative symptom scale (PANSS) and the Calgary Depression Scale for Schizophrenia (CDSS)
* Alcohol use disorder: Alcohol craving questionnaire self-report (ACQ-SR) and obsessive compulsive drinking scale (OCDS)
* Drug use disorders: Modified versions of the alcohol scales to make these relevant to the particular drug of abuse.
* Anorexia Nervosa: Yale-Brown-Cornell Eating Disorder Scale [YBC-EDS], Eating disorder examination questionnaire (EDE-Q)
* Bulimia Nervosa: Yale-Brown-Cornell Eating Disorder Scale [YBC-EDS], Eating disorder examination questionnaire (EDE-Q)
* Binge eating disorder: Young-Brown Obsessive Compulsive Scale Modified for Binge Eating [YBOCS-BE]
* OCD: Obsessive compulsive inventory (OCI) and Yale-Brown Obsessive Compulsive Scale (YBOCS)
* PTSD: Post-traumatic Stress Disorder Checklist-Civilian Version [PCL-C]
* Generalized anxiety disorder: Generalized Anxiety Disorder 7-item (GAD-7) scale
* Chronic pain: Numeric Rating Scale (NRS) for Chronic Pain
* Panic Disorder: Panic Disorder Severity Scale (PDSS)
* Somatoform Disorders: The Somatic Symptom Scale (SSS-8)
* Impulse Control disorders: Massachusetts General Hospital Hairpulling Scale (This questionnaire will be adapted depending on the urges the patient cannot control e.g. compulsive picking) BPD: The Borderline Evaluation of Severity Over Time (BEST)

At all time points, information regarding medication changes and other psychiatric treatments will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Received an intervention on the psychiatric inpatient unit at Stanford Hospital aimed at treating a major depressive episode or suicidal ideation

Exclusion Criteria:

-None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the psychiatric unit at Stanford University displaying depressive symptoms or suicidal ideation
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-07-09 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Montgomery-Asberg Depression Rating Scale (MADRS) | Weekly for first 4 weeks, followed by bi-weekly up until 24 weeks post-intervention
  This is a ten-item clinician rated questionnaire in which the clinician rates each item from 0-6. Scores of 6 indicate more severe depressive symptoms. Total scores are between 0 and 60 with scores >35 indicating severe depression. Response is defined as a 50% reduction or greater in MADRS score compared to baseline. Remission is defined as a MADRS score of <10.

SECONDARY OUTCOMES:
Scale for Suicide Ideation (SSI) | Weekly for first 4 weeks, followed by bi-weekly up until 24 weeks post-intervention
  Clinical assessment measuring suicidal thoughts & behaviors
Beck Depression Inventory II (BDI-II) | Weekly for first 4 weeks, followed by bi-weekly up until 24 weeks post-intervention
  The Beck Depression Inventory (BDI-II) is a 21-item, self-report rating inventory that measures characteristic attitudes and symptoms of depression. BDI-II items are rated on a 4-point scale ranging from 0 to 3 based on severity of each item. The maximum total score is 63.
  Scores: 0-13= minimal depression, 14-19=mild depression, 20-28=moderate depression, 29-63=severe depression
Columbia-Suicide Severity Rating Scale (C-SSRS) | Weekly for first 4 weeks, followed by bi-weekly up until 24 weeks post-intervention
  Self-report questionnaire identifying the presence or absence of six suicidal thoughts or behaviors in the past month or since the last visit. Each 'yes' answer is scored as 1, meaning the maximum total score is 6.
  The scale identifies specific behaviors which may be indicative of a person's intent to complete suicide. An person exhibiting even a single behavior identified by the scale was 8 to 10 times more likely to complete suicide.
Young Mania Rating Scale (YMRS) | Weekly for first 4 weeks, followed by bi-weekly up until 8 weeks post-intervention.
  11-item multiple choice clinician-rated questionnaire. Each question is rated from 0 to 4 with 4
Pittsburgh Insomnia Rating Scale (PIRS-20) | Weekly for first 4 weeks, followed by bi-weekly up until 8 weeks post-intervention.
  Self-report insomnia rating scale
Hamilton Rating Scale for Depression Six Item (HAMD-6) | Weekly for first 4 weeks, followed by bi-weekly up until 8 weeks post-intervention.
  Response is defined as a 50% reduction or greater in HAMD-6 score compared to baseline. HAMD-6 is a 6-item clinical assessment measuring depressive symptoms (scores range from 0-24 with scores of 5 or more indicating clinical levels of depression). The number of weeks in which HAMD-6 scores are lower than 50% of baseline will be calculated to provide a measure of duration of response.
Quick Inventory Depressive Symptomatology (QIDS) | Weekly for first 4 weeks, followed by bi-weekly up until 8 weeks post-intervention.
  Self-report measure of depressive symptoms
Immediate Mood Scaler (IMS-12) | weekly for first 4 weeks, followed by bi-weekly up until 8 weeks post-intervention.
  12-item self-report questionnaire used to measure current mood
Number of hospital re-admissions and service use | Bi-weekly up until 24 weeks post-intervention
  The number of times patients are re-admitted to hospital and used psychiatric services since the last assessment will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Nolan Williams, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford Hospital, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kelly MS, Oliveira-Maia AJ, Bernstein M, Stern AP, Press DZ, Pascual-Leone A, Boes AD. Initial Response to Transcranial Magnetic Stimulation Treatment for Depression Predicts Subsequent Response. J Neuropsychiatry Clin Neurosci. 2017 Spring;29(2):179-182. doi: 10.1176/appi.neuropsych.16100181. Epub 2016 Nov 30. PMID 27899052
- [Background] Haq AU, Sitzmann AF, Goldman ML, Maixner DF, Mickey BJ. Response of depression to electroconvulsive therapy: a meta-analysis of clinical predictors. J Clin Psychiatry. 2015 Oct;76(10):1374-84. doi: 10.4088/JCP.14r09528. PMID 26528644
- [Background] Berggren A, Gustafson L, Hoglund P, Johanson A. A long-term follow-up of clinical response and regional cerebral blood flow changes in depressed patients treated with ECT. J Affect Disord. 2014;167:235-43. doi: 10.1016/j.jad.2014.06.005. Epub 2014 Jun 12. PMID 24997226
- [Background] Murrough JW, Perez AM, Pillemer S, Stern J, Parides MK, aan het Rot M, Collins KA, Mathew SJ, Charney DS, Iosifescu DV. Rapid and longer-term antidepressant effects of repeated ketamine infusions in treatment-resistant major depression. Biol Psychiatry. 2013 Aug 15;74(4):250-6. doi: 10.1016/j.biopsych.2012.06.022. Epub 2012 Jul 27. PMID 22840761
- [Background] Dell'osso B, D'Urso N, Castellano F, Ciabatti M, Altamura AC. Long-term efficacy after acute augmentative repetitive transcranial magnetic stimulation in bipolar depression: a 1-year follow-up study. J ECT. 2011 Jun;27(2):141-4. doi: 10.1097/YCT.0b013e3181f66601. PMID 20966770